CLINICAL TRIAL: NCT02089191
Title: Comparison of Pre-Lens Tear Film Stability With Daily Disposable Contact Lenses Using Ring Mire Projection
Brief Title: Tear Film Stability of DAILIES® AquaComfort Plus® Contact Lenses vs. MyDay® Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: M-14-006
Record Dates: First submitted 2014-03-14; First posted 2014-03-17 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Refractive Error
Keywords: DACP; DAILIES® AquaComfort Plus; Tear film stability; NIK-BUT
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DACP/MyDay (Other): Nelfilcon A contact lenses worn in Period 1, with stenfilcon A contact lenses in Period 2. Each product worn bilaterally for 12 hours over 1 day.
  Interventions: Device: Nelfilcon A contact lenses; Device: Stenfilcon A contact lenses
- MyDay/DACP (Other): Stenfilcon A contact lenses worn in Period 1, with nelfilcon A contact lenses in Period 2. Each product worn bilaterally for 12 hours over 1 day.
  Interventions: Device: Nelfilcon A contact lenses; Device: Stenfilcon A contact lenses

INTERVENTIONS:
Device: Nelfilcon A contact lenses
  Other Names: DAILIES® AquaComfort Plus®; DACP
Device: Stenfilcon A contact lenses
  Other Names: MyDay®

SUMMARY:
The purpose of this study is to evaluate tear film stability of DAILIES® AquaComfort Plus® (DACP) compared to MyDay® after 12 hours of lens wear.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an Informed Consent form;
* Adapted, current soft contact lens wearer;
* Required contact lens prescription within the power range specified in the protocol (+6.00 to -10.00 diopters (D));
* Cylinder ≤ -1.00 D in both eyes at Visit 1;
* Vision correctable to 0.1 logarithm of the Minimum Angle of Resolution (logMAR) or better in each eye at distance with pre-study lenses at Visit 1;
* Willing to wear study lenses up to 12 hours and attend all study visits;
* Able to be successfully fitted with study lenses;
* Unstable tear film with a NIK-BUT value below 13 seconds in either eye without lenses;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any ocular infection, inflammation, abnormality, or active disease that would contraindicate contact lens wear;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the Investigator;
* Use of artificial tears and rewetting drops during the study;
* Monocular (only 1 eye with functional vision) or fit with only 1 lens;
* Any abnormal ocular condition observed during Visit 1;
* History of herpetic keratitis, ocular surgery, or irregular cornea;
* Pregnant or lactating;
* Participation in any clinical study within 30 days of Visit 1;
* Current MyDay® or DAILIES® AquaComfort Plus® lens wearer;
* Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Affairs, Clinical Manager, Vision Care, Study Director — Alcon Research
Locations (1):
- Alcon Investigative Site, Jena, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 investigational site located in Germany.
Groups:
- DACP/MyDay: Nelfilcon A contact lenses worn in Period 1, followed by stenfilcon A contact lenses in Period 2
- MyDay/DACP: Stenfilcon A contact lenses worn in Period 1, followed by nelfilcon A contact lenses in Period 2
Period: Period 1, First 12 Hours
Arm/Group | DACP/MyDay | MyDay/DACP
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0
Period: Period 2, Second 12 Hours
Arm/Group | DACP/MyDay | MyDay/DACP
Started | 15 (One participant discontinued between Period 1 and Period 2 due to availability) | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis group includes all enrolled participants.
Groups:
- Overall: Nelfilcon A and stenfilcon A contact lenses worn for 12 hours each in Period 1 and 2 as randomized
Arm/Group | Overall
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (3.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 9
Region of Enrollment [Number; unit: participants]
  Germany | 31

OUTCOME MEASURES:

1. Primary Outcome: Mean Time Post-blink to 15% Distortion of the Projected Rings After 12 Hours of Lens Wear
Description: The participant blinked twice, then kept eye open. Circular images were projected onto tear film layer located on the surface of the contact lens. Measuring software automatically detected areas where the tear film destabilized after the blink. The time to 15% destabilization of the tear film was calculated. A longer time indicates a more stable tear film. The right eye was evaluated.
Time Frame: Day 1, Hour 12, each period
Population: This analysis population includes all randomized subjects who did not meet the critical deviation criteria as specified in the Deviations and Evaluability Plan.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- DACP: Nelfilcon A contact lenses
- MyDay: Stenfilcon A contact lenses
Arm/Group | DACP | MyDay
Number analyzed (Participants) | 31 | 30
seconds | 22.84 (3.299) | 22.87 (3.026)

2. Secondary Outcome: Mean Speed of Tear Film Break-up at 15 Seconds Post-blink After 12 Hours of Lens Wear
Description: The participant blinked twice, then kept eye open. Circular images were projected onto tear film layer located on the surface of the contact lens. Measuring software automatically detected areas where the tear film destabilized after the blink. The slope of the regression line (distorted areas vs. time) was calculated. A slower speed (higher number) indicates a more stable tear film. The right eye was evaluated.
Time Frame: Hour 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent distortion per second
Arm/Group | DACP | MyDay
Number analyzed (Participants) | 31 | 30
percent distortion per second | 0.3 (0.38) | 0.2 (0.23)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (March 2014 to April 2014). This analysis population includes all participants/eyes exposed to any investigational product evaluated in this study.
Description: An adverse event was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical sign in subjects, users or other persons, whether or not related to the medical device.
Arm/Group | DACP | MyDay
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30

LIMITATIONS AND CAVEATS:
There was a high censoring rate observed with the objective measurements and therefore there are limitations to the conclusions that may be drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.